CLINICAL TRIAL: NCT00761605
Title: An Open-label Prospective, Non-comparative Study to Evaluate the Subjective Experiences Upon Transition to Paliperidone Extended Release(ER) in Subjects With Schizophrenia
Brief Title: Phase 4 Study to Evaluate Efficacy of Paliperidone Extended-Release(ER) in Schizophrenic Participants
Acronym: PASS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR015253; PAL-KOR-4003
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Results first posted 2014-03-06 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Paliperidone extended-release; Antipsychotics Agents
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paliperidone (Experimental): Paliperidone oral tablet will be administered once daily at a dose of 6 milligram (mg) for 24 weeks, wherein dose range was 3 to 12 mg per day.
  Interventions: Drug: Paliperidone

INTERVENTIONS:
Drug: Paliperidone — Paliperidone oral tablet will be administered once daily at a dose of 6 milligram (mg) for 24 weeks, wherein dose range was 3 to 12 mg per day.
  Other Names: R076477; Invega Extended-release tablet

SUMMARY:
The purpose of this study is to investigate the efficacy of flexibly dosed paliperidone extended-release (mechanism to dissolve a drug over time in order to be released slower and steadier into the blood stream) in improving or maintaining the subjective symptoms of the participants in three participants' groups (that is, by the reason to switch: lack of efficacy group, lack of tolerability group, and lack of compliance group) who switched from other previous antipsychotic drugs to paliperidone extended-release tablets at flexible doses.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), prospective (study following participants forward in time), single arm, and non-comparative study of paliperidone Extended-release (ER) in participants switching from the previous oral antipsychotic to flexibly dosed paliperidone ER. The total study duration will be approximately of 24 weeks per participant. The study consists of 2 parts: Screening (that is, 14 days before study commences on Day 1); Treatment (24 weeks). Efficacy will primarily be evaluated by change from baseline in symptom checklist 90-R (SCL90-R) at Week 24. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Childbearing potential women who consent to the use of the consistently permissible contraception (oral contraceptive, contraceptive injection, intrauterine device, double barrier method and contraceptive patch)
* Participants who are compliant with self-medication or can receive consistent help or support
* Participants who need to change the antipsychotic drug to another one for the following reasons among the participants treated with an antipsychotic drug for more than two weeks before the screening (1) Group of lack of efficacy: The antipsychotic drug is clinically required to be changed because there is no or little therapeutic response despite the appropriately dosed antipsychotic therapy (2) Group of lack of tolerance: The antipsychotic drug is required to be changed due to lack of tolerance to the existing antipsychotic drug or the safety issue (3) Group of lack of compliance: The antipsychotic drug is required to be changed due to lack of medication compliance or the participant wants to change the antipsychotic drug)

Exclusion Criteria:

* Participants with the past history of neuroleptic malignant syndrome (NMS)
* Participants who are suspicious of having clinically significant risk including suicide or aggressive behavior and are expected to unable to complete the study (based on the investigator's judgment)
* Participants with severe preexisting gastrointestinal narrowing (pathologic or iatrogenic) or participants who cannot swallow the drug whole (The study drug must not be chewed, divided, melted or grinded because it can impact the study drug release profile
* Female participants who are pregnant or are breast feeding
* Participants who have participated in any investigational drug trial within 1 month prior to the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2008-04; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea
Locations (8):
- South Korea (8):
  - Chunchun
  - Incheon
  - Inchun
  - Kangwondo
  - Kyunggido
  - Kyungki
  - Kyunki
  - Seoul

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone: Paliperidone oral tablet was administered once daily at a dose of 6 milligram (mg) for 24 weeks, wherein dose range was 3 to 12 mg per day.
Period: Overall Study
Arm/Group | Paliperidone
Started | 387
Completed | 246
Not Completed | 141
Not completed — Adverse Event | 26
Not completed — Death | 2
Not completed — Lack of Efficacy | 26
Not completed — Lost to Follow-up | 29
Not completed — Withdrawal by Subject | 37
Not completed — Other | 21

BASELINE CHARACTERISTICS:
Arm/Group | Paliperidone
Number analyzed (Participants) | 387
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.73 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 214
  Male | 173

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Symptom Checklist 90-R (SCL90-R) at Week 24
Description: The SCL90-R (Derogatis, 1992) measures 9 domains, including somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism, which provides a global index of distress, the Global Severity Index (GSI). SCL-90-R includes 90 items rated on 5-point scale, ranging from 0 (not at all) to 4 (extremely). Total scale score range from 0 to 360. Higher scores indicate worsening of disease. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: Intent to treat (ITT) population for efficacy included all the participants who received paliperidone extended-release (ER) at least once and who had at least 1 post baseline efficacy assessment. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone (Lack of Efficacy Group): Paliperidone Extended-release (ER) tablet at a dose ranging from 3 to 12 milligram (mg) per day was given orally for 24 weeks as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of efficacy (switching of antipsychotic drug was clinically necessary because of no or insufficient response to treatment despite antipsychotic drug therapy at an adequate dose).
- Paliperidone (Lack of Tolerability Group): Paliperidone ER tablet at a dose ranging from 3 to 12 mg per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of tolerability (switching of antipsychotic drug was necessary due to lack of tolerability or safety problem in the existing antipsychotic drug).
- Paliperidone (Lack of Compliance Group): Paliperidone ER tablet at a dose ranging from 3 to 12 mg per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of compliance (switching of antipsychotic drug was necessary due to lack of compliance in the existing antipsychotic drug).
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 277 | 78 | 32
Units on a scale
  Baseline | 99.84 (70.35) | 73.03 (57.60) | 67.66 (58.86)
  Change at Week 24 | 13.09 (57.78) | 8.87 (33.17) | 10.50 (42.33)

2. Secondary Outcome: Change From Baseline in Total Personal and Social Performance (PSP) Score at Week 24
Description: The PSP scale assesses the degree of dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (1, absent to 6, very severe) in each of the 4 domains. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less or equal to 30, functioning so poorly as to require intensive supervision. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: The ITT population for efficacy included all the participants who received paliperidone extended-release (ER) at least once and who had at least 1 post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Paliperidone (Lack of Efficacy Group): Paliperidone ER tablet at a dose ranging from 3 to 12 milligram (mg) per day was given orally for 24 weeks as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of efficacy (switching of antipsychotic drug was clinically necessary because of no or insufficient response to treatment despite antipsychotic drug therapy at an adequate dose).
- Paliperidone (Lack of Compliance Group): Paliperidone ER tablet at a dose ranging from 3 to 12 mg per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of compliance (switching of antipsychotic drug was necessary due to lack of tolerability or safety problem in the existing antipsychotic drug).
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 277 | 78 | 32
Units on a scale
  Baseline | 56.03 (15.51) | 63.62 (11.76) | 63.44 (16.07)
  Change at Week 24 | -5.81 (11.73) | -3.77 (8.12) | -4.59 (11.32)

3. Secondary Outcome: Change From Baseline in Subjective Well-being Under Neuroleptic (SWN-20) Scale at Week 24
Description: The SWN-20 scale is a 20 item scale that was originally designed to explore the subjective experience of psychotic participants. The SWN scale contains five sub-scales consisting of four items each: mental functioning (MF), self-control (SC), emotional regulation (ER), and social integration (SI), physical functioning (PF). The total score ranges from a minimum of 20 (poor subjective experience) to a maximum of 120 (excellent subjective experience). SWN scores appear to correlate with measure of objective psychopathology, quality of life and other self-ratings of mood. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: The ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment."N" (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 276 | 78 | 32
Units on a scale
  Baseline | 70.61 (17.09) | 76.67 (18.40) | 80.50 (17.01)
  Change at Week 24 | -1.54 (14.62) | -2.33 (15.11) | -1.06 (13.87)

4. Secondary Outcome: Change From Baseline in Sleep Quality Based on Visual Analog Scale at Week 24
Description: Sleep quality was assessed by an 11-point visual analog scale. Participants indicated on the 11-point visual analog scale (score ranging from 0 to 100 millimeter) how well they have slept in the previous 7 days, from 0 (very badly) to 100 (very well); and how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 100 (all the time). Scores were averaged for the previous 7 days. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 277 | 77 | 32
Millimeter (mm)
  Baseline | 65.62 (30.52) | 70.89 (24.90) | 62.45 (30.96)
  Change at Week 24 | 1.74 (36.00) | 3.66 (27.79) | -1.94 (34.18)

5. Secondary Outcome: Change From Baseline in Daytime Drowsiness Based on Visual Analog Scale at Week 24
Description: Daytime Drowsiness was assessed by an 11-point visual analog scale. Participants indicated on the 11-point visual analog scale (score ranging from 0 to 100 millimeter) how well they have slept in the previous 7 days, from 0 (very badly) to 100 (very well); and how often they have felt drowsy within the previous 7 days, from 0 (not at all) to 100 (all the time). Scores were averaged for the previous 7 days. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Millimeter (mm)
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 277 | 77 | 32
Millimeter (mm)
  Baseline | 43.27 (31.65) | 39.40 (28.02) | 44.47 (28.12)
  Change at Week 24 | 4.80 (33.31) | 2.42 (30.84) | 7.83 (36.24)

6. Secondary Outcome: Change From Baseline in Krawiecka Scale Score at Week 24
Description: Psychopathology of participants was assessed by Krawiecka scale. Psychopathology of participants was assessed by Krawiecka scale, score ranges from 0 to 16. Higher score indicates worsening of disease. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 277 | 78 | 32
Units on a scale
  Baseline | 5.38 (3.28) | 4.74 (2.99) | 4.38 (3.02)
  Change at Week 24 | 1.43 (2.62) | 1.32 (1.94) | 1.69 (2.72)

7. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Week 24
Description: The CGI-S rating scale is a 7 point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: ITT population for efficacy included all the participants who received paliperidone extended-release (ER) at least once and who had at least 1 post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 277 | 78 | 32
Units on a scale
  Baseline | 3.77 (1.16) | 3.46 (0.98) | 3.25 (1.05)
  Change at Week 24 | 0.70 (1.04) | 0.47 (0.86) | 0.47 (0.95)

8. Secondary Outcome: Change From Baseline in Clinical Global Impression - Improvement (CGI-I) Score at Week 24
Description: The CGI-I is a 7-point scale that requires the clinician to assess how much the participant's illness has improved or worsened relative to a baseline state at the beginning of the intervention and rated as: 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Change from Baseline was calculated as value at Baseline minus value at Week 24. Data for three groups is presented here, based on participants' transition to Paliperidone ER from other oral antipsychotics.
Time Frame: Baseline and Week 24
Population: The ITT population for efficacy included all the participants who received paliperidone extended-release (ER) at least once and who had at least 1 post baseline efficacy assessment. "N" (number of participants analyzed) signifies participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Paliperidone (Lack of Efficacy Group) | Paliperidone (Lack of Tolerability Group) | Paliperidone (Lack of Compliance Group)
Number analyzed (Participants) | 268 | 76 | 31
Units on a scale
  Baseline | 3.63 (0.91) | 3.66 (0.60) | 3.48 (1.00)
  Change at Week 24 | 0.46 (1.23) | 0.37 (0.96) | 0.35 (1.17)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 24
Description: Safety population included all the eligible participants who received paliperidone extended-release (ER) at least once .
Arm/Group | Paliperidone
Serious Adverse Events (participants affected / at risk) | 38/387
Other Adverse Events (participants affected / at risk) | 209/387
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone (N=387)
Acute myocardial infarction (Cardiac disorders) | 1
Hyperprolactinaemia (Endocrine disorders) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Colon cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Acute psychosis (Psychiatric disorders) | 1
Aggression (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 5
Delusion (Psychiatric disorders) | 3
Hallucination (Psychiatric disorders) | 2
Hallucination, auditory (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 1
Panic attack (Psychiatric disorders) | 1
Psychiatric symptom (Psychiatric disorders) | 1
Psychotic disorder (Psychiatric disorders) | 7
Schizophrenia (Psychiatric disorders) | 5
Suicide attempt (Psychiatric disorders) | 3
Cholecystectomy (Surgical and medical procedures) | 1
Gastrectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone (N=387)
Hyperprolactinaemia (Endocrine disorders) | 8
Oculogyration (Eye disorders) | 8
Constipation (Gastrointestinal disorders) | 13
Nausea (Gastrointestinal disorders) | 11
Nasopharyngitis (Infections and infestations) | 9
Weight decreased (Investigations) | 10
Weight increased (Investigations) | 36
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 15
Akathisia (Nervous system disorders) | 44
Bradykinesia (Nervous system disorders) | 9
Dizziness (Nervous system disorders) | 16
Extrapyramidal disorder (Nervous system disorders) | 8
Headache (Nervous system disorders) | 33
Sedation (Nervous system disorders) | 10
Somnolence (Nervous system disorders) | 20
Tremor (Nervous system disorders) | 23
Anxiety (Psychiatric disorders) | 22
Depression (Psychiatric disorders) | 11
Hallucination, auditory (Psychiatric disorders) | 8
Insomnia (Psychiatric disorders) | 48
Amenorrhoea (Reproductive system and breast disorders) | 15

LIMITATIONS AND CAVEATS:
Some Adverse Events summaries were reported based on estimates due to the fact that they were not prepared in the original study report and the relevant definitions of the data elements were not available for these summaries to be regenerated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less